CLINICAL TRIAL: NCT05620862
Title: Phase I Dose Escalation and Pharmacokinetics Clinical Trial of Mitoxantrone Hydrochloride Liposome in Children With Relapsed and Refractory Lymphoma and Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yizhuo Zhang, Director, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-Ly -K01
Record Dates: First submitted 2022-11-08; First posted 2022-11-17 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Pediatric Solid Tumor
MeSH Terms: interventions — Irinotecan; Vincristine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mitoxantrone hydrochloride liposome alone or combined with Irinotecan+Vincristine (Experimental): In phase Ia, patients with relapsed and refractory lymphoma and solid tumors will receive mitoxantrone hydrochloride liposome alone (at three doses of 16 mg/m2, 20 mg/m2 and 24 mg/m2, ) or combination of Irinotecan 50mg/ m2，d1-5, Vincristine 1.5mg/ m2，d1 for up to 6 cycles (21 days per cycle). In phase Ib, patients will recive mitoxantrone hydrochloride liposome 24 mg/m2, combination of Irinotecan 50mg/ m2，d1-5, Vincristine 1.5mg/ m2
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome; Drug: Irinotecan; Drug: Vincristine

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome — In phase Ia, mitoxantrone hydrochloride liposome will be administered by an intravenous infusion at three doses of 16 mg/m2, 20 mg/m2 and 24 mg/m2 . In phase Ib, mitoxantrone hydrochloride liposome will be administered by an intravenous infusion of 24mg/m2. Up to 6 cycles (21 days per cycle)
Drug: Irinotecan — 50mg/ m2，d1-5, 21 days per cycle
Drug: Vincristine — Vincristine 1.5mg/ m2，d1 , 21 days per cycle

SUMMARY:
Phase I dose escalation clinical trial: to explore the dose limiting toxicity (DLT) of mitoxantrone hydrochloride liposome injection in the treatment of children with relapsed and refractory lymphoma and solid tumors.

Pharmacokinetics clinical trial: to observe the pharmacokinetics of mitoxantrone hydrochloride liposomes in children with relapsed and refractory lymphoma and solid tumors.

To evaluate the safety and efficacy of mitoxantrone hydrochloride liposomes in children with lymphoma and solid tumors.

DETAILED DESCRIPTION:
This is a phase I dose escalation and pharmacokinetics clinical trial to evaluate the safety and efficacy of mitoxantrone hydrochloride liposomes in children with lymphoma and solid tumors. In the phase Ia dose escalation study, patients with relapsed and refractory lymphoma and solid tumors will be treated with mitoxantrone hydrochloride liposome alone or combined treatment at the dose of 16 mg/m2, 20 mg/m2 and 24 mg/m2, each cohort wil enroll 9~18 children. Simultaneously 6~15 cases were added for pharmacokinetic study to ensure 8 cases are included in each dose group with the same mitoxantrone hydrochloride liposome dose. In phase Ib, patients received the combination therapy of mitoxantrone hydrochloride liposome at the MTD dose (24mg/m2) .

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects fully understand and voluntarily participate in this study and sign the informed consent form (ICF);
* 2. 2-21 years old;
* 3. Expected survival ≥ 3 months;
* 4. Subjects with histologically confirmed diagnosis of relapsed and refractory lymphoma and solid tumors, which is one of the following subtypes:

  1. Lymphoblastic lymphoma
  2. Anaplastic large T cell lymphoma
  3. Burkitt's lymphoma
  4. Diffuse large B-cell lymphoma
  5. Peripheral T, NK/T cell lymphoma
  6. Soft tissue sarcoma
  7. Neuroblastoma
  8. Other subtypes of lymphoma or solid tumors that the investigators believe can be included
* 5. Relapsed lymphoma is defined as the lymphoma that relapse after obtaining complete response (CR) after initial chemotherapy; Refractory lymphoma subjects meet one of the following conditions: 1) The tumor shrinks <50% or disease progression after 4 cycles of standard chemotherapy,; 2) CR after standard chemotherapy, but relapse within half a year; 3) 2 or more relapses after CR; 4) relapse after hematopoietic stem cell transplantation;
* 6. Lymphoma subjects must have at least one evaluable or measurable lesion per lugano2014 criteria: for lymph node lesions, the length should be > 1.5cm; For non-lymph node lesions, the length should be > 1.0cm;
* 7. Solid tumors must have tumor lesions measurable by CT or MRI;
* 8. ECOG Performance Status: 0-2;
* 9. Bone marrow function: Absolute neutrophil count ≥1.5×109/L, Platelet count ≥75×109/L, Hemoglobin ≥ 80g/L (Absolute neutrophil can be relaxed to ≥ 1.0×109/L, Platelet count can be relaxed to ≥50×109/L, Hemoglobin can be relaxed to ≥75 g/L in subjects with poor bone-marrow reserve);
* 10. Liver and kidney function: serum creatinine ≤ 1.5×ULN (upper limit of normal); AST and ALT ≤ 2.5×ULN (≤ 5×ULN for subjects with liver metastases); total bilirubin ≤ 1.5×ULN (≤ 3×ULN for subjects with liver metastases).

Exclusion Criteria:

* 1. The subject had previously received any of the following anti-tumor treatments:

  1. Subjects who have been treated with mitoxantrone or mitoxantrone liposomes;
  2. Previously received doxorubicin or other anthracycline treatment, and the total cumulative dose of doxorubicin was more than 360 mg/m2 (1 mg doxorubicin equivalent to 2 mg epirubicin);
  3. Subjects who received anti-tumor treatment (including chemotherapy, targeted therapy, glucocorticoid, traditional Chinese medicine with anti-tumor activity, etc.) or participated in other clinical trials and received trial drugs;
  4. Subjects who received autologous hematopoietic stem cell transplantation within 100 days after the first medication or allogeneic hematopoietic stem cell transplantation.
* 2. Hypersensitivity to any study drug or its components;
* 3. Uncontrolled systemic diseases (such as active infection, uncontrolled hypertension, diabetes, etc.);
* 4. Heart function and disease meet one of the following conditions:

  1. Long QTc syndrome or QTc interval > 480 ms;
  2. Complete left bundle branch block, grade II or III atrioventricular block;
  3. Serious and uncontrolled arrhythmias requiring drug treatment;
  4. New York Heart Association grade ≥ III;
  5. Cardiac ejection fraction (LVEF)< 50%;
  6. A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.
* 5. Hepatitis B and hepatitis C active infection (plus HBV DNA if one positive for hepatitis B surface antigen or core antibody and HBV DNA more than 1×103 copy/mL excluded; plus HCV RNA if hepatitis C antibody positive and HCV RNA more than 1×103 copy/mL exclude);
* 6. Human immunodeficiency virus (HIV) infection (HIV antibody positive);
* 7. Subjects with other malignant tumors past or present (except for non-melanoma skin basal cell carcinoma, breast/cervical carcinoma in control, and other malignant tumors that have been effectively controlled without treatment within the past five years);
* 8. Subjects suffering from primary or secondary central nervous system (CNS) lymphoma or a history of CNS lymphoma at the time of recruitment;
* 9. Pregnant and lactating women and childbearing age patients unwilling to take contraceptive measures;
* 10. Unsuitable subjects for this study determined by the investigator.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose | Up to 21 days
  To investigate the safety and preliminary antitumor efficacy
peak time (Tmax) | Up to 18 weeks
  To evaluate the pharmacokinetics of mitoxantrone hydrochloride liposome at different doses in subjects
Maximum Plasma Concentration (Cmax) | Up to 18 weeks
  To evaluate the pharmacokinetics of mitoxantrone hydrochloride liposome at different doses in subjects
Area under the plasma concentration versus time curve (AUC) | Up to 18 weeks
  To evaluate the pharmacokinetics of mitoxantrone hydrochloride liposome at different doses in subjects
Elimination half life (t1/2) | Up to 18 weeks
  To evaluate the pharmacokinetics of mitoxantrone hydrochloride liposome at different doses in subjects
Incidence and severity of hematological adverse events | From date of randomization until 4 weeks after the last dose
  To evaluate the incidence and severity of hematological adverse events in patients enrolled in phase Ib

SECONDARY OUTCOMES:
Dose limiting toxicities | Up to 21 days
  To investigate the safety
Objective response rate | Up to 18 weeks
  To investigate the preliminary antitumor efficacy of phase I dose escalation and pharmacokinetics study
Complete response rate | Up to 18 weeks
  To investigate the preliminary antitumor efficacy of phase I dose escalation and pharmacokinetics study
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 70 weeks
  To investigate the preliminary antitumor efficacy of phase I dose escalation and pharmacokinetics study
The incidence and severity of AE and SAE | up to 42 weeks unless related serious adverse events need to be recorded indefinitely
  To identify the incidence and severity of AE and SAE (NCI CTCAE v5.0)
Incidence and severity of non-hematological adverse events | From date of randomization until 4 weeks after the last dose
  The incidence and severity of non-hematological adverse events were evaluated in patients enrolled in Phase Ib

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No